CLINICAL TRIAL: NCT02879994
Title: A Phase II Study of Pembrolizumab in EGFR Mutant, Tyrosine Kinase Inhibitor Naïve Treatment Patients With Advanced Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Pembrolizumab in Treating Patients With EGFR Mutant, Tyrosine Kinase Inhibitor Naive Advanced Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-001818; NCI-2016-00861 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); Garon Pembrolizumab IST NSCLC; 15-001818 (Other: UCLA / Jonsson Comprehensive Cancer Center)
Record Dates: First submitted 2016-08-23; First posted 2016-08-26 (Estimated); Results first posted 2021-07-14 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2019-09

CONDITIONS: Stage IIIA Non-Small Cell Lung Cancer; Stage IIIB Non-Small Cell Lung Cancer; Stage IV Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (pembrolizumab) (Experimental): Patients receive pembrolizumab IV over 30 minutes on day 1. Treatment repeats every 3 weeks for up to 35 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Pembrolizumab

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475

SUMMARY:
This phase II trial studies how well pembrolizumab works in treating patients with epidermal growth factor receptor (EGFR) mutant non-small cell lung cancer that have not received prior tyrosine kinase inhibitor therapy and has spread to other places in the body. Monoclonal antibodies, such as pembrolizumab, may block growth in different ways by targeting certain cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine efficacy (objective response rate (ORR)) of front-line pembrolizumab for metastatic EGFR mutation positive programmed cell death 1 ligand 1 (PD-L1)+ (> 1% by immunohistochemistry [IHC]) non-small cell lung cancer (NSCLC).

SECONDARY OBJECTIVES:

I. Determine safety (adverse event tabulation and grading) of front-line pembrolizumab for metastatic EGFR mutation positive PD-L1+ (> 1% by IHC) NSCLC.

II. Determine efficacy (progression free survival (PFS), overall survival (OS)) of front-line pembrolizumab for metastatic EGFR mutation positive PD-L1+ (>1% by IHC) NSCLC.

III. Determine ORR, PFS and OS of subsequent EGFR tyrosine kinase inhibitor (TKI) therapy in patients with EGFR-sensitizing mutation after pembrolizumab.

TERTIARY OBJECTIVE:

I. Analyze tumor tissue biomarkers for potential correlation with response.

OUTLINE:

Patients receive pembrolizumab intravenously (IV) over 30 minutes on day 1. Treatment repeats every 3 weeks for up to 35 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for up at 3 and 6 months, and then every 9 weeks thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information (PHI)
* Have a life expectancy of at least 3 months
* Have a histologically or cytologically confirmed diagnosis of non-small cell lung cancer (NSCLC) and have at least one measurable lesion as defined by modified Response Evaluation Criteria in Solid Tumors (RECIST) 1.1; the target lesion(s) should also have bi-dimensional measurability for RECIST 1.1 evaluation on study
* Have an EGFR mutation (sensitizing or non-sensitizing)
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) performance scale
* Absolute neutrophil count (ANC) >= 1,500 /microliters(mcL)
* Platelets >= 100,000 / mcL
* Hemoglobin >= 9 g/dL or >= 5.6 mmol/L without transfusion or erythropoietin (EPO) dependency (within 7 days of assessment)
* Serum creatinine =< 1.5 X upper limit of normal (ULN) OR measured or calculated creatinine clearance (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance (CrCl)) >= 60 mL/min for subject with creatinine levels > 1.5 x institutional ULN
* Serum total bilirubin =< 1.5 x ULN OR direct bilirubin =< ULN for subjects with total bilirubin levels > 1.5 ULN
* Aspartate transaminase (AST) (serum glutamic oxaloacetic transaminase (SGOT)) and alanine transferase (ALT) (serum glutamate pyruvate transaminase (SGPT)) =< 2.5 X ULN OR =< 5 X ULN for subjects with liver metastases
* Albumin >= 2.5 mg/dL
* International Normalized Ratio (INR) or Prothrombin Time (PT) =< 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants
* Activated partial thromboplastin time (aPTT) =< 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
* Have provided tissue for PD-L1 biomarker analysis from a newly obtained formalin fixed tumor tissue from a biopsy of a tumor lesion not previously irradiated; the tissue sample must be received and evaluated by the study site prior to start of treatment; fine needle aspirates are not acceptable; needle or excisional biopsies, or resected tissue is required
* Have a PD-L1 positive (either strongly or weakly) tumor as determined by the IHC 22C3 pharmDx test at the study site; if a patient's initial tumor specimen is not classified as PD-L1 positive by the central laboratory, a newly obtained specimen (different from the sample previously submitted) may be submitted for testing; if the newer specimen is classified as PD-L1 positive by the study site, the patient meets this eligibility criterion
* Have resolution of toxic effect(s) of the most recent prior chemotherapy to grade 1 or less (except alopecia); if subject received major surgery or radiation therapy of > 30 Gy, they must have recovered from the toxicity and/or complications from the intervention
* Female subject of childbearing potential has a negative urine or serum pregnancy test; if the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required; the serum pregnancy test must be negative for the subject to be eligible
* Female subjects may be enrolled in the trial if they are:

  * of non-childbearing potential which is defined as:
  * of childbearing potential who are willing to use either 2 adequate barrier methods or a barrier method plus a hormonal method of contraception to prevent pregnancy, or to abstain from heterosexual activity throughout the trial, starting with the screening visit (visit 1) through 120 days after the last dose of MK-3475 (pembrolizumab)
* Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy

Exclusion Criteria:

* Has received prior therapy with an EGFR tyrosine kinase inhibitor (such as erlotinib, gefitinib, afatinib, rociletinib, or AZD9291) for NSCLC
* Is currently participating or has participated in a study of an investigational agent or using an investigational device within 30 days of the first dose of trial treatment; the 30 day window should be applied to the last dose of an antineoplastic investigational agent or last use of an investigational device with antineoplastic intent
* Is receiving systemic steroid therapy within three days prior to the first dose of trial treatment or receiving any other form of immunosuppressive medication (corticosteroid use on study for management of early combined immunosuppression (ECIs) is allowed)
* Is expected to require any other form of systemic or localized antineoplastic therapy while on trial (including maintenance therapy with another agent for NSCLC or radiation therapy)
* Has received prior systemic cytotoxic chemotherapy, antineoplastic biological therapy (e.g., cetuximab), major surgery within 3 weeks of the first dose of trial treatment; received thoracic radiation therapy of > 30 Gy within 6 months of the first dose of trial treatment
* Has received prior therapy with an anti-programmed cell death protein 1 (PD-1), anti-PD-L1, anti-programmed cell death 1 ligand 2 (PD-L2), anti-cluster of differentiation 137 (CD137), or anti-cytotoxic t-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways); has participated in another MK-3475 clinical trial
* Has a known history of prior malignancy except if the patient has undergone potentially curative therapy with no evidence of that disease recurrence for 3 years since initiation of that therapy; Note: the time requirement for no evidence of disease for 3 years does not apply to the NSCLC tumor for which a subject is enrolled in this trial; the time requirement also does not apply to subjects who underwent successful definitive resection of basal cell carcinoma of the skin, superficial bladder cancer, squamous cell carcinoma of the skin, or in situ cervical cancer
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis; subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by magnetic resonance imaging [MRI] for at least two weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are using no steroids for at least three days prior to study medication
* Has an active autoimmune disease, or a documented history of autoimmune disease that required systemic steroids or immunosuppressive agents; subjects with vitiligo or resolved childhood asthma/atopy would be exception to this rule; subjects that require inhaled steroid or local steroid injections will not be excluded from the study; subjects with hypothyroidism not from autoimmune disease and stable on hormone replacement will not be excluded from the study
* Has had an allogeneic tissue/solid organ transplant
* Has interstitial lung disease or a history of pneumonitis that required oral or intravenous glucocorticoids to assist with management; lymphangitic spread of the NSCLC is not exclusionary
* Has received or will receive a live vaccine within 30 days prior to the first administration of study medication; seasonal flu vaccines that do not contain live virus are permitted
* Has an active infection requiring intravenous systemic therapy
* Has known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies)
* Has known active hepatitis B or C; active hepatitis B is defined as a known positive hepatitis B surface antigen (HBsAg) result; active hepatitis C is defined by a known positive hepatitis (Hep) C antibody (Ab) result and known quantitative hepatitis C virus (HCV) ribonucleic acid (RNA) results greater than the lower limits of detection of the assay
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Is, at the time of signing informed consent, a regular user (including "recreational use") of any illicit drugs or had a recent history (within the last year) of substance abuse (including alcohol)
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit (visit 1) through 120 days after the last dose of MK-3475

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-09-15 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2019-01-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward Garon, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States

REFERENCES:
- [Derived] Lisberg A, Cummings A, Goldman JW, Bornazyan K, Reese N, Wang T, Coluzzi P, Ledezma B, Mendenhall M, Hunt J, Wolf B, Jones B, Madrigal J, Horton J, Spiegel M, Carroll J, Gukasyan J, Williams T, Sauer L, Wells C, Hardy A, Linares P, Lim C, Ma L, Adame C, Garon EB. A Phase II Study of Pembrolizumab in EGFR-Mutant, PD-L1+, Tyrosine Kinase Inhibitor Naive Patients With Advanced NSCLC. J Thorac Oncol. 2018 Aug;13(8):1138-1145. doi: 10.1016/j.jtho.2018.03.035. Epub 2018 Jun 1. PMID 29874546

RESULTS

PARTICIPANT FLOW:
Recruitment Details: September 15, 2016 - October 24, 2018 Recruitment Period
Period: Overall Study
Arm/Group | Treatment (Pembrolizumab)
Started | 11
Completed | 0
Not Completed | 11
Not completed — off treatment early | 7
Not completed — Adverse Event | 2
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Population: Male and female subjects with EGFR mutant, tyrosine kinase inhibitor naïve, PD-L1+, advanced non-small cell lung cancer
Arm/Group | Treatment (Pembrolizumab)
Number analyzed (Participants) | 11
Age, Customized [Count of Participants; unit: Participants]
  18 - 21 years | 0
  22 - 29 years | 0
  30 - 39 years | 1
  40 - 49 years | 0
  50 - 59 years | 3
  60 - 69 years | 6
  70 - 79 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) Determined as the Percentage of Patients Achieving Complete Response or Partial Response as Respectively Defined in RECIST 1.1
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by accessed by radiographic imaging: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to 14 months
Population: Enrollment was ceased due to lack of efficacy after 11 of 25 planned patients were treated. Only 1 patient had an objective response, but repeat analysis of this patient's tumor definitively showed the original report of an epidermal growth factor receptor (EGFR) mutation to be erroneous.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Pembrolizumab)
Number analyzed (Participants) | 11
Participants | 1

2. Secondary Outcome: Number of Participants With Adverse Events According to the National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0
Description: Number of Participants with Adverse Events According to the National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0
Time Frame: Up to 14 Months
Population: Enrollment was halted after 11 of 25 planned subjects due to lack of efficacy.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Pembrolizumab)
Number analyzed (Participants) | 11
Participants | 11

3. Secondary Outcome: Efficacy (Progression Free Survival (PFS) and Overall Survival (OS)) Assessed by RECIST 1.1
Description: Will evaluate Progression Free Survival and Overall Survival. Average of Progression Free Survival recorded for limited number of subjects analyzed. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: assessed for up to 14 months
Population: Participants analyzed is 10 because although 11 patients were treated, forensic analysis revealed that 1 subject did not have documented EGFR mutation. Regarding Overall Survival, median OS was not reached at time of data cutoff.
Measure: Mean (Full Range); unit: days
Arm/Group | Treatment (Pembrolizumab)
Number analyzed (Participants) | 10
days
  Progression free survival | 119 [42 to 123]
  Overall Survival: number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 14 months
Description: Period of active patient enrollment
Arm/Group | Treatment (Pembrolizumab)
All-Cause Mortality (participants affected / at risk) | 2/11
Serious Adverse Events (participants affected / at risk) | 6/11
Other Adverse Events (participants affected / at risk) | 6/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Pembrolizumab) (N=11)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypotension (Metabolism and nutrition disorders) | 1 (1)
Hypercalcemia (Blood and lymphatic system disorders) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Elevated alanine aminotransferase (Hepatobiliary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Pembrolizumab) (N=11)
Rash (Skin and subcutaneous tissue disorders) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Adrenal insufficiency (Endocrine disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Flu-like symptoms (General disorders) | 2 (2)
Chills (General disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Hyperglycemia (Gastrointestinal disorders) | 1 (1)
Anorexia (Psychiatric disorders) | 1 (1)
Alanine aminotransferase increased (Blood and lymphatic system disorders) | 1 (1)
Aspartate aminotransferase increased (Blood and lymphatic system disorders) | 1 (1)
Thyroid-stimulating hormone decreased (Blood and lymphatic system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-12-01): https://cdn.clinicaltrials.gov/large-docs/94/NCT02879994/Prot_SAP_000.pdf
  • Informed Consent Form (2018-02-14): https://cdn.clinicaltrials.gov/large-docs/94/NCT02879994/ICF_001.pdf